CLINICAL TRIAL: NCT06854679
Title: A Feasibility Study in Dose Escalated Treatment in Rectal Cancer on Mr-Linac Using Mr GuidED Adaptive Radiotherapy
Brief Title: Dose Escalated Radiotherapy for Rectal Cancers Using MR-guided Radiotherapy
Acronym: ANDROMEDA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR 5774
Record Dates: First submitted 2024-12-03; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-12

CONDITIONS: Rectal Adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiotherapy dose escalation (Experimental): All patients will receive 45Gy in 25# to mesorectum and elective nodal volumes, and 52.5Gy in 25# as standard to primary gross tumour volume which includes primary tumour, visible nodal disease and extramural vascular invasion if present. Boost dose escalation to a maximum of 60Gy will be delivered to patients with ongoing visible disease from week 2 of treatment onwards.
  Interventions: Radiation: Radiotherapy dose escalation

INTERVENTIONS:
Radiation: Radiotherapy dose escalation — All patients will receive 45Gy in 25# to mesorectum and elective nodal volumes, and 52.5Gy in 25# as standard to primary gross tumour volume which includes primary tumour, visible nodal disease and extramural vascular invasion if present. Boost dose escalation to a maximum of 60Gy will be delivered to patients with ongoing visible disease from week 2 of treatment onwards.

SUMMARY:
Standard radiotherapy in the UK involves having daily chemotherapy tablets with radiotherapy treatment for 5 weeks at a dose of 52.5Gy to the rectal cancer over 25 fractions. This is the likely treatment participants will be having if they decide not to take part in this study. Increasing the dose to 60Gy is shown to increase the chance that rectal cancer will be treated completely, a term known as "complete pathological response". Patients who have a complete pathological response after their treatment can avoid surgery and enter into a surveillance programme to monitor for early signs of the cancer returning. Surveillance can mean 3-6 months camera tests and MRI scans depending on the local unit. If these patients continue to show signs of complete pathological response then they can avoid long term complications from surgery such as a stoma. Unit studies have shown that that increasing the dose of radiotherapy can cause slightly more bowel and bladder side effects, but using adaptive radiotherapy to limit radiotherapy to normal tissue could keep the rate of bothersome side effects as low, which is similar as standard treatment.

All adaptive treatments within this trial will be delivered on a state of the art, radiotherapy machine called an MR-linac (Magnetic Resonance Linear Accelerator). It combines an MRI scanner with a radiotherapy treatment machine called a Linear Accelerator (called a 'linac' for short). The use of the MR-linac means there is no extra radiation dose given when taking daily images to check for the position of participants rectal cancer (unlike CT scans or X-ray). It also enables the investigators to adapt or 'tweak' the radiotherapy plan each day to match the exact position of the rectal cancer and adjacent organs. The non-adaptive fractions can be delivered on either the MR-Linac or CT-linac depending on factors such as treatment machine availability.

The investigators will deliver the treatment on the MR-linac using a technique called intensity modulated radiotherapy (precise X-ray treatment, called IMRT for short). IMRT is able to mould radiotherapy treatment according to what the investigators can see, therefore enabling the investigators to give highly targeted treatment. The investigators already have considerable experience in delivering radiotherapy to rectal cancer with this machine and now wish to focus on whether they could increase dose to benefit long term outcome for all rectal cancer patients as well as reducing the side effects of treatment.

The purpose of this research is to increase the dose to rectal cancer while adapting to the changes that the investigators can see to the rectal cancer during treatment. This means that if the rectal cancer is seen to reduce in size they will be able to deliver a 'shrinking boost' according to what can be seen. This will enable the investigators to give high dose radiotherapy to the cancer whilst limiting radiotherapy to healthy tissue. Without the ability to adapt to changes that the investigators see to the tumour throughout the entire treatment course, standard treatment delivers dose to a larger area of surrounding healthy tissue to ensure that the tumour is sufficiently targeted.

The investigators want to find out if by using this adaptive, shrinking boost approach, they can safely increase radiotherapy dose to rectal cancer, whilst limiting the side effects you experience, in comparison with standard treatment. If this is possible, then this would lead into further clinical trial where the investigators would compare outcomes of higher-dose treatment to standard-of-care. The investigators can't be certain that the side effects will be different, and they don't know if this treatment results in the best chance of cancer cure. However they know from other studies that this is the likely outcome, with surgery being delayed for patients. Patients who have a complete pathological response after combined chemotherapy and radiotherapy treatment enter into a surveillance programme where MRI and camera tests (flexible sigmoidoscopy) are performed at regular intervals looking for early signs of cancer returning.

The investigators expect that the chance of participants having a complete pathological response with this technique is higher than with standard dose, although the investigators can't know this for sure until they have completed further studies. It is possible that the cure rate may be lower or higher than the standard dose.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged ≥18 years
* Histological confirmation of locally advanced rectal adenocarcinoma requiring neoadjuvant chemoradiotherapy as per RMH clinical guidelines.
* Patients suitable for concomitant chemotherapy
* Patients with disease included within treatment field size of MR-Linac.
* WHO Performance status 0-2
* Ability of the participant understand and the willingness to sign a written informed consent form.
* Ability/willingness to comply with the patient reported outcome questionnaires schedule throughout the study.

Exclusion Criteria:

* Contraindications to MRI (e.g. pacemaker, potentially mobile metal implant, claustrophobia)
* Disease outside maximum radiotherapy treatment field length.
* Comorbidities which predispose to significant toxicity (e.g. inflammatory bowel disease) or preclude long term follow up
* Unilateral or bilateral total hip replacement, or other pelvic metalwork which causes artefact on diffusion-weighted imaging
* Previous pelvic radiotherapy
* Patients needing induction chemotherapy prior to chemoradiotherapy
* Previous invasive malignancy within the last 2 years excluding basal or squamous cell carcinomas of the skin, low risk non-muscle invasive bladder cancer (assuming cystoscopic follow up now negative) or small renal masses on surveillance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2027-01-13 (Estimated); Study Completion 2029-01-13 (Estimated)

PRIMARY OUTCOMES:
Number of patients completing 90% or more fractions delivered on MR-Linac. | Up to 12 weeks
  To establish the technical feasibility of delivering adaptive dose escalated radiotherapy on an MR-Linac.

SECONDARY OUTCOMES:
• Physician reported gastrointestinal (GI) and genitourinary (GU) toxicity (CTCAE grade) at baseline and the end of treatment then at 6 and 12 weeks post-treatment. | 24 months post completing treatment
  • Physician reported gastrointestinal (GI) and genitourinary (GU) toxicity (CTCAE grade) at baseline and the end of treatment then at 6 and 12 weeks post-treatment.
• Late toxicity (CTCAE) at 1 and 2 years post-treatment. | 24 months post completing treatment
  • Late toxicity (CTCAE) at 1 and 2 years post-treatment.
• Recurrence/progression assessment for up to 2 years following completion of treatment. | 24 months post completing treatment
  • Recurrence/progression assessment for up to 2 years following completion of treatment.
• Post-treatment pathological response assessment at 6 weeks with MRI using Mandard response grading. If complete pathological response on MRI then patient will undergo surgical surveillance with sigmoidoscopy and biopsy. If ongoing disease patient will | 24 months post completing treatment
  • Post-treatment pathological response assessment at 6 weeks with MRI using Mandard response grading. If complete pathological response on MRI then patient will undergo surgical surveillance with sigmoidoscopy and biopsy. If ongoing disease patient will have appropriate surgical technique for removal of tumour.
• Patient-reported outcome measures (PROMs) | 24 months post completing treatment
  Patient-reported outcome measures (PROMs) from the QLQ-CR29 and QLQ-C30 questionnaires. Patients will be asked to complete PROMs at 6 and 12 weeks, 6 months, 1 and 2 years post treatment. Scale of 1(low impact) to 4 (high impact)

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden Hospital, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided